CLINICAL TRIAL: NCT01846676
Title: Assessment of the "Active Communication Education" Program for Audiological Rehabilitation in Patients With Hearing Loss Users of Hearing Aids
Brief Title: Assessment of the ACE Program for Rehabilitation in Hearing Loss
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Chile (Other)
Responsible Party: Principal Investigator, Felipe Cardemil, Otolaryngology department, University of Chile, University of Chile
Allocation: Non-Randomized | Model: Single Group | Masking: Triple | Purpose: Treatment
Other Study IDs: 221-2010
Record Dates: First submitted 2013-04-29; First posted 2013-05-03 (Estimated); Last update posted 2017-01-13 (Estimated); Status verified 2017-01

CONDITIONS: Hearing Loss
Keywords: Hearing loss, rehabilitation programs, adherence to hearing aids.
MeSH Terms: conditions — Hearing Loss

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Program counseling (Active Comparator): Active branch, subject to the rehabilitation program
  Interventions: Behavioral: Active Communication Education Program
- No counseling (Placebo Comparator): Passive branch, which was control, with usual management (no intervention).
  Interventions: Other: Control

INTERVENTIONS:
Behavioral: Active Communication Education Program — The program called Active Communication Education (ACE), that is a semistructured rehabilitation program for people with hearing loss, which aims to improve rehabilitation of hearing aids users by a strategy based on problem solution.
  Arms: Program counseling
Other: Control — Participants in this arm will not receive intervention during the study protocol time. After the completion of the protocol, they will receive the same intervention that the intervention group, meaning the ACE program intervention.
  Arms: No counseling

SUMMARY:
* Introduction: Hearing loss is a prevalent condition in elderly population. However, the low adherence to hearing aids is a fact, with an estimation of use of 50 per cent. In 2007 there was designed a rehabilitation program called ACE, which aims to improve rehabilitation directed to hearing aids users. The study hypothesis is that a counseling program will improve adherence to hearing aids in elderly population.
* Objective: To evaluate the utility of a standardized counselling program in patients with hearing loss.
* Material and Methods: A before/after trial will be carried out, approved by the Hospital ethics - committee. Patients with 65 years and older with hearing loss diagnosed by pure tone audiometry will be included. To assess adherence we will use the IOI-HA scale.

DETAILED DESCRIPTION:
* Introduction: Hearing loss is a prevalent condition in elderly population. However, the low adherence to hearing aids is a fact, with an estimation of use of 50 per cent. In Chile, hearing aids are provided by the State for elderly population. In 2007 there was designed a rehabilitation program called Active Communication Education (ACE), that is a semistructured rehabilitation program for people with hearing loss, which aims to improve rehabilitation of hearing aids users by a strategy based on problem solution.
* The study hypothesis is that a counseling program will improve adherence to hearing aids in elderly population.
* Objective: To evaluate the utility of a standardized counseling program in patients with hearing loss.
* Material and Methods: A before/after clinical trial will be carried out, approved by the Hospital ethics - committee. Patients with 65 years and older diagnosed by pure tone audiometry who are beneficiaries of the Public GES hearing loss programme and receive a hearing aid will be included. The subjects will be randomized in two branches: Active branch, subject to the rehabilitation program; and passive branch, which was control, with usual management (no intervention). To assess adherence we will use the IOI-HA scale.

ELIGIBILITY:
Inclusion Criteria:

* Bilateral hearing loss equal or higher than 40 decibels
* Age 65 years old or more
* Agree to be included in the study
* Have a relative to go to the intervention with the subject

Exclusion Criteria:

* Severe organic brain impairment
* Physical or mental incapacity to understand the study questionnaires
* Structural pathology of the ear that produces hearing loss as chronic otitis media, ear canal tumor, or tumor of the cerebellopontine angle

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 180 (Actual)
Dates: Start 2012-10; Primary Completion 2013-10 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Adherence to the use of hearing aids in elderly population with hearing loss | One year

CONTACTS AND LOCATIONS:
Overall Officials: Felipe Cardemil, MD, Principal Investigator — University of Chile
Locations (1):
- Barros Luco Trudeau Hospital, San Miguel, Santiago, Santiago Metropolitan, Chile